CLINICAL TRIAL: NCT07067723
Title: Epidemiological and Clinical Characteristics of Human Mpox Outbreak in Equateur Province in the Democratic Republic of Congo (Part3)
Brief Title: Epidemiological and Clinical Characteristics of Human Mpox Outbreak in Equateur Province in the Democratic Republic of Congo (Part2)
Status: Enrolling by invitation | Type: Observational
Sponsor: Osaka Metropolitan University (Other)
Responsible Party: Principal Investigator, Yasutoshi KIDO, Professor, Osaka Metropolitan University
Other Study IDs: N553/BN/PMMF/2024-2
Record Dates: First submitted 2025-05-14; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Monkeypox (Mpox)
Keywords: contact tracing; transmission; outbreak investigation
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin lesion and oral mucosa swab sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is

* to better understand the dominant modes of transmission
* to estimate the extent of transmission among contacts by determining the secondary infection rate for human-to-human transmission at an individual level and identifying factors associated with secondary infections.
* to determine the proportion of asymptomatic or pauci-symptomatic infections.
* to characterize the incubation period of mpox and the duration of infectiousness, including reproduction numbers.
* to assess serological responses following confirmed infection.

DETAILED DESCRIPTION:
Mpox is caused by the monkeypox virus (MPXV), a member of the genus Orthopoxvirus (family Poxviridae). This virus is closely related to the variola virus, which causes smallpox. MPXV was first identified in 1958, and the first human case was reported in the Democratic Republic of the Congo (DRC) in 1970. It was presumed that the smallpox (vaccinia) vaccine would confer cross-protection against mpox. Following the global eradication of smallpox in 1980, mpox remained largely confined to limited regions in Central Africa-where zoonotic spillover from wild animal reservoirs constituted the primary route of transmission. Equateur Province is among the areas in the DRC with a notably high burden of reported mpox cases.

Over the past five decades, routine smallpox vaccination ceased worldwide, resulting in waning herd immunity against orthopoxviruses. During this period, mpox incidence rose markedly, with an estimated tenfold increase in global cases. Two principal genetic clades of MPXV have been identified: clade I (historically referred to as the Congo Basin clade) and clade II (the West African clade). In 2018, Nigeria experienced a resurgence of mpox, highlighting the virus's potential to emerge in previously controlled areas. Starting in 2022, clade II mpox circulated globally, especially among men who have sex with men (MSM), peaking in mid-2022 before declining to persistently lower levels by early 2023. Although clade II mpox typically exhibits a low case-fatality ratio (<1%), clade I has historically been associated with more severe disease and higher mortality. In 2023, the number of reported mpox cases continued to climb in the DRC, prompting the World Health Organization (WHO) to declare a Public Health Emergency of International Concern (PHEIC) in August 2024.

Recent surveillance indicates that sub-clade Ia MPXV is spreading in western DRC through multiple transmission modes, including contact with infected wild animals, household exposure, or sexual contact. By contrast, sub-clade Ib mpox in the eastern part of the country appears initially to spread via intimate or sexual contact between adults, followed by household transmission. Numerous environmental and social risk factors-including the consumption of rodent species, deforestation, climate change, civil unrest, population displacement, emerging MPXV variants, and weakened immunity-may be driving mpox incidence. Clade Ia mpox is currently affecting western parts of the DRC, yet the epidemiology remains poorly understood due to the limited number of laboratory-confirmed cases.

This study aims to better understand the dominant modes of transmission of Mpox in Equateur Province in DRC and to estimate the extent of transmission among contacts by determining the secondary infection rate for human-to-human transmission at an indicidual level and identifying factors associated with secondary infections. The findings will advance understanding of mpox transmission dynamics, ultimately informing more effective prevention and control strategies in endemic settings.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent:

Proxy-assisted informed consent is allowed under safety considerations. Following oral consent, the investigator will document this on the informed consent form as a witness.

Fulfillment of the current mpox clinical case definition in the DRC, which includes:

Presence of a vesicular or pustular eruption with deep-seated, firm pustules.

At least one of the following symptoms:

Fever preceding the eruption. Lymphadenopathy (inguinal, axillary, or cervical). Presence of pustules or crusts on the palms of the hands or soles of the feet.

Laboratory confirmation:

At least one molecular-based mpox diagnostic test confirming the diagnosis.

Exclusion Criteria:

* Participants will be excluded from the study under the following conditions:

Refusal to participate in the study:

Individuals who decline to provide consent for study participation will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study targets laboratory-confirmed cases of mpox and their contacts, defined based on exposure to the primary case within the household or in external settings (e.g., workplaces, social interactions).
  This study targets patients reported as suspected mpox cases (all ages, both sexes) to the Health District Central Office in the selected sites. The study population is designed to minimize selection bias related to health-seeking behavior.
  Cases are defined as Individuals who reported to local health agents with symptoms consistent with mpox and subsequently tested positive for mpox through a molecular-based diagnostic test.
  Contacts are defined as individuals identified as having close contact with a laboratory-confirmed mpox case. Close contact includes but is not limited to the following type of contact.
Sampling Method: Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Transmission chain | through study completion, average 4 weeks
  Definition: The sequence and structure of mpox transmission events within households and beyond, including identification of primary and secondary cases.
  To map transmission dynamics and determine how mpox spreads within close-contact settings. Detailed epidemiological tracing and genetic sequencing to confirm transmission links.
Incubation Period | through study completion, an average 4 weeks
  Definition: The time between exposure to the mpox virus and the onset of symptoms.
  To estimate the range and median incubation period of mpox based on detailed exposure history and symptom onset data. Exposure dates and symptom onset dates from confirmed cases and their contacts.
Serial Interval | through study completion, an average 4 weeks
  Definition: The time between the onset of symptoms in a primary case and the onset of symptoms in a secondary case they infect.
  To estimate the serial interval of mpox, which is critical for understanding transmission timelines and epidemic control. Symptom onset dates for linked cases within households and other close-contact settings.
Secondary Attack Rate (SAR) | through study completion, an average 4 weeks
  Definition: The proportion of susceptible household contacts who develop mpox after exposure to a confirmed case.
  To quantify transmission efficiency within households and identify risk factors influencing SAR.
Effective Reproduction Number (Re) | through study completion, an average of 2 years
  Definition: The average number of secondary cases generated by a single infectious individual in the current population.
  To estimate Re during the study period, which reflects real-time transmission potential under existing control measures. Based on observed transmission chains and SAR data.

CONTACTS AND LOCATIONS:
Overall Officials: Yasutoshi Kido, Professor, Principal Investigator — Osaka Metropolitan University
Locations (1):
- Equateur Provincial Public Health Laboratory, Mbandaka, Équateur Province, Democratic Republic of the Congo